CLINICAL TRIAL: NCT02435264
Title: Assessing the Barriers and Motivators to Providing and Consuming Healthier Foods in the Singaporean Hawker Center Setting and Evaluating the Healthier Hawker Programme (Now Called the Healthier Dining Program)
Brief Title: Choosing Healthier Eating Options at Work and School
Acronym: Project CHEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rob M van Dam (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Sponsor-Investigator, Rob M van Dam, Associate Professor, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11-137
Record Dates: First submitted 2015-04-21; First posted 2015-05-06 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Healthier Food Consumption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthier Dining Program Intervention (Experimental): Food centers that receive the Healthier Dining Program (HDP)
  Interventions: Other: Healthier Dining Program Intervention
- Control centers (No Intervention): Food centers that do not receive the Healthier Dining Program (HDP)

INTERVENTIONS:
Other: Healthier Dining Program Intervention — The food environment at the intervention centers will be modified to increase the availability of healthier foods and low calorie meals.
  Arms: Healthier Dining Program Intervention

SUMMARY:
Recent national statistics revealed that the prevalence of lifestyle related diseases is increasing in Singapore. Much of this disease burden can be prevented using lifestyle strategies. A large proportion of Singaporeans consume foods prepared by outside vendors. These foods are typically high in refined-grains and saturated fat, and choices for healthier foods like brown-rice often do not exist. The Healthier Dining Program managed by the Health Promotion Board of Singapore, seeks to assess if increasing the availability of healthier food options increases consumer consumption of these foods. The investigators aim to evaluate this program implemented on the National University of Singapore campus. A major output of this evaluation will be the assessment of the barriers and enablers to programme implementation which will provide guidance for the widespread implementation of the programme. Additionally this evaluation can lead to detailed recommendations on policies and programmes relevant to non-home food environments. This is important as successful interventions have the potential of improving the eating behaviors of a vast majority of the population.

DETAILED DESCRIPTION:
The evaluation will use a cluster randomized controlled design in 3 test NUS eateries with 3 control eateries that are matched on type (canteen or food court) and on similarity of students/staff that it typically serves (example: consumers from arts or sciences faculties). It will include both process evaluation and outcome evaluation components. The primary purpose of the process evaluation will be to understand the enablers or barriers to programme implementation which will help to adjust the programme as it is being implemented and to assess whether the intervention elements are being implemented as planned. The primary purpose of the outcome evaluation will be to assess if healthier options are available and if consumers are buying these healthier options. The investigators will triangulate data sources and use both quantitative and qualitative data to inform this evaluation.

Specific aims include

1. To conduct a process evaluation of the Healthier Dining Program (HDP) by assessing the reach, fidelity, dose delivered, dose received, and by examining the contextual barriers and facilitators towards the Healthier Dining Program implementation at NUS
2. To assess the effects of the HDP on the knowledge, attitudes, and behavior of hawkers and consumers regarding healthier food options
3. To conduct a cost effectiveness evaluation of the HDP
4. To model the impact of changes in dietary intakes ascribed to the HDP intervention, on the incidence of type-2 diabetes and cardiovascular diseases in Singapore using statistical modeling and computer simulation

A total of 408 consumers at baseline and 10 weeks after the intervention (68 persons per cluster, 34 staff and 34 students) will be interviewed. The sample size was computed based on a proportion difference of 40 % (5 % in the control centers and 45% in the intervention centers) of consumers who eat healthier foods at least once per week. Healthier foods include wholegrain foods, less sugar/ healthier choice symbol (HCS) beverage and reduced calorie meals, foods that are being targeted by the programme. A power of 0.8,a two-sided alpha of 0.05, an intra-cluster correlation of 0.15, and a drop-out rate of 25 % for consumers was assumed. Centers will be matched based on type (canteen or food court) and on similarity of students/staff that it typically serves (example; consumers from arts or sciences faculties) and will be randomized to either the intervention or control group. All eligible and consenting hawkers at the NUS canteens and food courts in the study will interviewed (approximately 15 per center, for a total of 90 hawkers).

ELIGIBILITY:
Inclusion Criteria:

* Food vendors:

  21 years or older Must be stall owner or decision maker
* Consumers 18 year or older (NUS students) or 21 years or older Frequent consumers of foods at NUS canteens or foodcourts

Exclusion criteria:

* Consumers:
* Persons unlikely to be on campus during the follow-up interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Changes in proportion of participants consuming healthier meals | Baseline, 10 weeks post intervention
  We will compare the between-arm difference in proportion of participants who had healthier meals prepared from out-of-home sources at least once a week at the post-intervention time-point.
  This information is based on data collected using a 7-day food diary. This is a well established method of dietary assessment. Diary information was reviewed in-person or via phone calls by trained researchers and processed via an in-house food composition database called E-Food system.
  Each meal consumed by the participant was assessed for whether it was prepared using either the healthier oil blends (≤ 35% saturated fat), wholegrain rice, low-sodium salt, or was lower in calorie (<500 kcal per serving). A meal that had at least one of these intervention-related characteristics was deemed as being a healthier meal. We will also conduct this analysis separately for each specific healthy meal type.

SECONDARY OUTCOMES:
Differences in out-of-home dietary intake of key nutrients | Baseline, 10 weeks post intervention
  We will assess the difference in dietary intakes of key nutrients from out-of-home meals between intervention and control arms. Specifically we will look at differences in consumption (g/1000 kcal) of monounsaturated fat, polyunsaturated fat, saturated fat, total fat and fibre, and the ratio of polyunsaturated fat to saturated fat. These key nutrients are likely to be modified by the intervention.
  This information is based on data collected using a 7-day food diary. This is a well established method of dietary assessment. Diary information was reviewed in-person or via phone calls by trained researchers before being processed through an in-house food composition database called E-Food system. The system used food composition data from the Singapore's Health Promotion Board FOCOS food composition database and U.S. Department of Agriculture (USDA) Nutrient Database for Standard Reference.
Differences in total dietary intake of key food groups | Baseline, 10 weeks post intervention
  We will assess the difference in total (out of home and home prepared) dietary intakes of key food groups between intervention and control arms. These include fruits,vegetables, snacks (savoury, sweet), rice (brown, white), noodles (regular, wholegrain), breads (regular, wholegrain) and beverages ( unsweetened, less sweet, regular)
  A short 20-question food frequency questionnaire (FFQ), derived from Singapore National Nutrition Survey 2010 was used to collect this information. Participants were asked to choose from four categories of intake frequencies ('per day', 'per week', 'per month' and 'never') for a serving of the food or beverage item over the month preceding the interview. Number of servings of these foods groups consumed on a weekly basis were calculated from this information.

IPD SHARING:
Plan to Share IPD: No